CLINICAL TRIAL: NCT00002765
Title: PHASE I STUDY OF ANTI-TAC(Fv)-PE38 (LMB-2), A RECOMBINANT SINGLE-CHAIN IMMUNOTOXIN FOR TREATMENT OF TAC-EXPRESSING MALIGNANCIES
Brief Title: Immunotoxin in Treating Patients With Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064729; NCI-96-C-0064F; NCI-T95-0042N; NCT00001501 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-05-06 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2003-03

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; Waldenström macroglobulinemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; prolymphocytic leukemia; recurrent mantle cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — B3(Fv)-PE38KDEL recombinant immunotoxin

INTERVENTIONS:
Biological: LMB-2 immunotoxin

SUMMARY:
RATIONALE: Immunotoxins can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of LMB-2 immunotoxin in treating patients who have leukemia or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the therapeutic efficacy and toxicity of the recombinant immunotoxin LMB-2, an anti-Tac murine monoclonal antibody fragment conjugated to a truncated portion of Pseudomonas exotoxin, in patients with Tac-expressing leukemias and lymphomas.
* Define the pharmacokinetics of LMB-2, including the terminal elimination serum half-life, area under the curve, and volume of distribution.
* Evaluate, in a preliminary manner, the immunogenicity of LMB-2 in these patients.
* Determine the effect of LMB-2 on various components of the circulating cellular immune system.

OUTLINE: This is a dose escalation study.

Patients receive LMB-2 immunotoxin IV over 30 minutes on days 1, 3, and 5. Treatment repeats every 15-21 days for up to 10 courses in the absence of disease progression, neutralizing antibodies, or unacceptable toxicity.

Cohorts of 3-6 patients each receive escalating doses of LMB-2 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 patient experiences dose limiting toxicity.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's disease, non-Hodgkin's lymphoma, or leukemia in one of the following categories:

  * Adult T-cell leukemia or lymphoma (ATL)

    * No smoldering ATL
    * No limitation on prior therapy
  * Cutaneous T-cell lymphoma (CTCL)

    * Stages IB-III and failed at least 1 standard therapy
    * Stage IV regardless of prior therapy
  * Stages I-IV peripheral T-cell lymphoma

    * Relapsed after standard chemotherapy
    * Ineligible for or refused salvage chemotherapy or bone marrow transplantation (BMT)
  * B-cell non-Hodgkin's lymphoma (NHL) of any histology

    * Indolent stages II-IV NHL

      * Failed at least 1 standard therapy
      * Disease symptomatic and requiring treatment
    * Aggressive NHL

      * Relapsed after standard chemotherapy
      * Ineligible for or refused salvage chemotherapy or BMT
  * Chronic lymphocytic leukemia (CLL)

    * Rai stages III and IV or Binet stage C
    * Failed standard therapy and at least 1 salvage chemotherapy
  * Primary B-cell prolymphocytic leukemia or prolymphocytic transformation of CLL

    * Failed standard therapy and at least 1 salvage chemotherapy
  * Hairy cell leukemia

    * Failed standard and salvage chemotherapy
    * Ineligible for or refused further salvage chemotherapy or BMT
  * Acute myelogenous leukemia

    * Failed standard chemotherapy
    * Ineligible for or refused salvage chemotherapy or BMT
  * Stages II-IV Hodgkin's disease

    * Failed standard chemotherapy
    * Ineligible for curative salvage radiotherapy or chemotherapy
    * Ineligible for or refused BMT
  * Patients with leukemias or lymphomas not easily classified in above categories who have failed standard therapy and are ineligible for or have refused bone marrow transplant
* Evidence of interleukin-2 receptor-alpha (IL2Ra) expression by one of the following:

  * Greater than 10% of malignant cells reactive with anti-Tac by immunohistochemistry
  * Greater than 10% of malignant cells from a particular site positive by FACS
  * Greater than 400 IL2Ra sites per malignant cell by radiolabeled anti-Tac binding
  * Soluble IL2Ra level greater than 1,000 U/mL (normal geometric mean 235, with 95% confidence levels of 112-502 U)
  * Hodgkin's disease with measurable disease not amenable to biopsy
* No CNS disease requiring treatment

  * Malignant cells in CSF allowed if judged not to represent clinically significant leukemic or lymphomatous meningitis (as in CSF contamination by blood)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* Greater than 2 months

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm3*
* Platelet count greater than 50,000/mm3* NOTE: *nonleukemic patients

Hepatic:

* AST and ALT less than 5 times normal

Renal:

* Creatinine less than 2.0 mg/dL OR
* Creatinine clearance greater than 50 mL/min

Pulmonary:

* FEV1, TLC, and DLCO greater than 50% of predicted if pulmonary or mediastinal involvement with tumor greater than one third of total thoracic diameter

Other:

* HIV negative
* Not pregnant
* Fertile patients must use effective contraception
* Serum must neutralize no more than 75% LMB-2 in tissue culture

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 3 weeks since prior interferon

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior cytotoxic chemotherapy
* At least 3 weeks since prior retinoids
* No concurrent chemotherapy

Endocrine therapy:

* No concurrent corticosteroids unless begun at least 3 weeks prior to entry and dose not increased during 3 weeks prior to entry

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior whole-body electron beam radiotherapy
* Other radiotherapy allowed within 3 weeks of entry provided less than 10% of marrow irradiated and measurable disease exists outside radiation port

Surgery:

* Not specified

Other:

* See Disease Characteristics
* At least 3 weeks since any prior systemic therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-04

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Laboratory of Molecular Biology, Bethesda, Maryland
  - Medicine Branch, Bethesda, Maryland

REFERENCES:
- [Background] Matsushita K, Margulies I, Onda M, Nagata S, Stetler-Stevenson M, Kreitman RJ. Soluble CD22 as a tumor marker for hairy cell leukemia. Blood. 2008 Sep 15;112(6):2272-7. doi: 10.1182/blood-2008-01-131987. Epub 2008 Jul 2. PMID 18596230
- [Background] Kreitman RJ, Margulies I, Stetler-Stevenson M, Wang QC, FitzGerald DJ, Pastan I. Cytotoxic activity of disulfide-stabilized recombinant immunotoxin RFB4(dsFv)-PE38 (BL22) toward fresh malignant cells from patients with B-cell leukemias. Clin Cancer Res. 2000 Apr;6(4):1476-87. PMID 10778980
- [Background] Robbins DH, Margulies I, Stetler-Stevenson M, Kreitman RJ. Hairy cell leukemia, a B-cell neoplasm that is particularly sensitive to the cytotoxic effect of anti-Tac(Fv)-PE38 (LMB-2). Clin Cancer Res. 2000 Feb;6(2):693-700. PMID 10690555
- [Result] Kreitman RJ, Wilson WH, White JD, Stetler-Stevenson M, Jaffe ES, Giardina S, Waldmann TA, Pastan I. Phase I trial of recombinant immunotoxin anti-Tac(Fv)-PE38 (LMB-2) in patients with hematologic malignancies. J Clin Oncol. 2000 Apr;18(8):1622-36. doi: 10.1200/JCO.2000.18.8.1622. PMID 10764422
- [Result] Kreitman RJ, Wilson WH, Robbins D, Margulies I, Stetler-Stevenson M, Waldmann TA, Pastan I. Responses in refractory hairy cell leukemia to a recombinant immunotoxin. Blood. 1999 Nov 15;94(10):3340-8. PMID 10552943